CLINICAL TRIAL: NCT06620848
Title: A Study of HRS-4642 Monotherapy or in Combination With Adebrelimab in Patients With Advanced Biliary Tract Tumors.
Brief Title: A Study of HRS-4642 Monotherapy or in Combination With Adebrelimab in the Treatment of Advanced Biliary Tract Tumors.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jia Fan, M.D, Shanghai Zhongshan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTC-2nd-IIT-HRS4642-SHR1316
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer
Keywords: KRAS G12D; Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HRS-4642 monotherapy arm (Experimental): Patients will receive HRS-4642 monotherapy at a fixed dose.
  Interventions: Drug: HRS-4642 monotherapy
- combination therapy arm (Experimental): Patients will receive HRS-4642 and adebrelimab combination therapy.
  Interventions: Drug: HRS-4642 and adebrelimab combination therapy

INTERVENTIONS:
Drug: HRS-4642 monotherapy — HRS-4642 will be administrated per dose level in which the patients are assigned.
  Arms: HRS-4642 monotherapy arm
Drug: HRS-4642 and adebrelimab combination therapy — HRS-4642 and adebrelimab will be administrated per dose level in which the patients are assigned.
  Arms: combination therapy arm

SUMMARY:
The study was designed to evaluate the efficacy and safety of HRS-4642 monotherapy or in combination with adebrelimab in the treatment of advanced biliary tract tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female.
2. Histologically or cytologically confirmed diagnosis of advanced biliary tract cancer.
3. Unresectable or metastatic advanced patients with progression or intolerance for ≥ one line of systemic therapy, including patients who metastasize during or within 6 months after neoadjuvant or adjuvant therapy (adjuvant therapy or neoadjuvant therapy must include gemcitabine-based chemotherapy).
4. Have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
5. ECOG performance status of 0-1.
6. With a life expectancy of ≥3 months.
7. Have adequate laboratory parameters and organ functions during the screening period.

Exclusion Criteria:

1. Known history of hypersensitivity to any components of HRS-4642 or adebrelimab.
2. Prior anti-tumor chemotherapy within 4 weeks before the study drug administration. Small molecular targeted drugs (including oral targeted drugs for other clinical trials) with a half-life of less than 5 or 7 days from the first medication.
3. Patients with untreated or active central nervous system tumor metastasis.
4. Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST V1.1 | up 2 years
  The ORR is defined as complete remission (CR) rate + partial remission (PR) rate by RECIST V1.1.
Adverse events(AEs), serious adverse events（SAEs） | up 2 years
  AEs and SAEs occurred from the first dose of treatment to 30 days after the last dose of HRS-4642 or 90 days after the last dose of adebrelimab (whichever comes late).

SECONDARY OUTCOMES:
Disease control rate (DCR) | up 2 years
  The DCR is defined as complete remission (CR) rate + partial remission (PR) rate + stable disease (SD).
Progression-free survival (PFS) | up 2 years
  PFS is defined as Time from the date of enrollment to of disease
Overall survival (OS) | up 2 years
  OS is defined as time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, M.D, Principal Investigator — Shanghai Zhongshan Hospital; Guoming Shi, M.D, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No